CLINICAL TRIAL: NCT00952458
Title: Bispectral Index Monitoring as an Adjunct to Standard Monitoring of Sedation During Endoscopic Retrograde Cholangiopancreaticography
Brief Title: Bispectral Index Monitoring of Sedation During Endoscopic Retrograde Cholangiopancreaticography
Acronym: EndoBISs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: II. Medizinische Klinik, Dr. Stefan von Delius, Klinikum rechts der Isar der Technischen Universität München
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2094/08
Record Dates: First submitted 2009-08-02; First posted 2009-08-06 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2010-05

CONDITIONS: Gastrointestinal Endoscopy; Sedation
Keywords: Safety; Midazolam and propofol sedation; ERCP; Bispectral Index monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIS monitoring (Experimental): Dosing of sedatives with BIS monitoring
  Interventions: Device: BIS monitoring
- Standard monitoring (No Intervention): Dosing of sedatives without BIS monitoring

INTERVENTIONS:
Device: BIS monitoring — Neuromonitoring of depth of sedation with Bispectral Index
  Arms: BIS monitoring

SUMMARY:
This randomized study investigates the benefits of an additional Bispectral Index monitoring of depth of sedation during endoscopic retrograde cholangiopancreaticography. A bispectral index (BIS) monitor is a neurophysiological monitoring device which continually analyses a patient's electroencephalograms during general anaesthesia to assess the level of consciousness during anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Indication for ERCP (Endoscopic Retrograde Cholangiopancreatography) with midazolam and propofol sedation

Exclusion Criteria:

* Missing informed consent
* ASA V
* Preexisting neurological deficit
* Known pregnancy
* Hypotension (RRsys<90mmHg), bradycardia (HR<50/min), hypoxia (SaO2<90%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary complications of sedation | 1-4 hours

SECONDARY OUTCOMES:
Efficacy of sedation | 1-4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stefan von Delius, MD, Principal Investigator — Klinikum rechts der Isar der Technischen Universität München
Locations (1):
- Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Background] von Delius S, Thies P, Rieder T, Wagenpfeil S, Herberich E, Karagianni A, Frimberger E, Meining A, Ludwig L, Ebert MP, Schulte-Frohlinde E, Neu B, Prinz C, Schmid RM, Huber W. Auditory evoked potentials compared with bispectral index for monitoring of midazolam and propofol sedation during colonoscopy. Am J Gastroenterol. 2009 Feb;104(2):318-25. doi: 10.1038/ajg.2008.73. Epub 2009 Jan 20. PMID 19190608